CLINICAL TRIAL: NCT05298306
Title: A Two-part Proof-of-Concept Study Assessing the Safety and Efficacy of LAT8881 in Lumbar Radicular Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lateral Pharma Pty Ltd (Industry)
Collaborators: Southern Star Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAT-NP-002
Record Dates: First submitted 2022-03-03; First posted 2022-03-28 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Radiculopathy Lumbar

STUDY DESIGN:
Intervention Model Description: The crossover study (Part B) is preceded by a single ascending dose study (Part A)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LAT8881 (Experimental): In Part A, LAT8881 will be given as a single intravenous infusion on separate days at doses of 0.8, 1.2 and 1.8 mg/kg.
  In Part B, LAT8881 will be given as a single intravenous infusion. The dose will be determined from the results of Part A.
  Interventions: Drug: LAT8881
- Placebo (Placebo Comparator): Matching placebo will be given as a single intravenous infusion in Part A and Part B
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LAT8881 — In Part A, LAT8881 will be given as a single intravenous infusion at doses of 0.8, 1.2 and 1.8 mg/kg.
  In Part B, a single intravenous infusion of LAT8881 will be given, the dose to be determined by the results in Part A
  Arms: LAT8881
Drug: Placebo — Matching placebo'given as a single intravenous infusion at all dose levels
  Arms: Placebo

SUMMARY:
The study consists of two parts. Part A will evaluate the safety and tolerability of intravenous LAT8881 in healthy volunteers using an ascending dose schedule. Part B will evaluate the analgesic efficacy of a single intravenous dose of LAT8881, compared with placebo, in patients with lumbar radicular pain.

Healthy volunteers are not accepted for Part B.

DETAILED DESCRIPTION:
Part A of this study is a double-blind, randomized, placebo-controlled, single ascending dose study of intravenous administration of LAT8881 over 5 minutes in healthy volunteers. Each participant has three treatment days, 1 infusion per dosing day, on Days 1, 4 and 7 as well as two short visits for safety blood sampling on Days 3 and 6. Subjects in Part A are randomized to receive placebo and LAT8881 according to the following treatment sequences. Two subjects are allocated to each treatment sequence, a total of eight subjects overall.

0.8 mg/kg/1.2 mg/kg/1.8 mg/kg;

0.8 mg/kg/1.2 mg/kg/Placebo;

0.8 mg/kg/Placebo/1.8 mg/kg;

Placebo/1.2 mg/kg/1.8 mg/kg.

Part B of this study is is a placebo-controlled randomized double blind cross-over safety and efficacy study of LAT8881 in up to 20 patients with lumbar radicular pain. Participants will be randomly assigned to one of two groups, to receive either LAT8881 then placebo or placebo then LAT8881. Participants will receive either a single dose of LAT8881 [the Maximum Tolerated Dose from Part A of the study] or placebo via intravenous administration over 5 minutes on two consecutive days.

ELIGIBILITY:
Key Inclusion Criteria:

For PART A, the following inclusion criteria apply:

* Male or female healthy participants, aged 18-49 years inclusive at screening;
* Body mass index of ≥ 19.0 kg/m2 to ≤ 32.0 kg/m2 at screening;
* Female participants must not be pregnant or breastfeeding
* Male participants with a female partner of childbearing potential must use highly effective contraception for 60 days after the last dose of study treatment

For PART B, the following key inclusion criteria apply:

* Male or female participants with unilateral pain, aged 18 years and above at screening;
* Body mass index of ≥ 19.0 kg/m2 at screening.
* Female participants must not be pregnant or breastfeeding
* Male participants with a female partner of childbearing potential must use highly effective contraception for 60 days after the last dose of study treatment
* Presenting with a history of unilateral pain, radiating into a lower limb, of lancinating, burning, stabbing or electric quality, of duration of >3 months.
* Pain scores (NRS) for average daily leg pain at rest at the relevant nerve root of a mean of ≥4/10 and ≤9/10 for 3 days prior to treatment, with a minimum of >3/10 on any day.
* Demonstration of disc herniation within 6 months by CT or MRI at a segmental level consistent with the clinical features.
* The site of disc herniation must affect L1-2, L2-3, L3-4, L4-5 or L5-S1.
* The patient is willing to keep all analgesic medication and other therapy usage stable or decreased in the week prior to, and a week after, IP administration.
* The patient is in good general health, with the exception of the presenting condition under study

Key Exclusion Criteria:

The following key exclusion criteria apply for both PART A and PART B:

* Any condition which might be a risk to participant safety or interfere with study evaluation
* Unwillingness to abstain from alcohol or nicotine products as required

The following additional key exclusion criteria apply to PART B:

* A history of significant pain unrelated to disc herniation that would significantly compromise assessment of leg radicular pain.
* Radiological evidence of foraminal stenosis or of clinically significant spinal stenosis .
* Lumbar back surgery related to the specific disc.
* Injection of an epidural corticosteroid injection within 3 months of screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Ludbrook, MBBS, Principal Investigator — Royal Adelaide Hospital
Locations (1):
- PARC Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in two parts. Part A was a single ascending dose study of intravenous LAT8881 in healthy volunteers. The second part of the study (Part B) was initiated after completion of Part A and was a crossover study of LAT8881 in subjects with lumbar radicular pain. Both parts of the study were randomized, placebo-controlled and double-blinded.
Pre-assignment Details: Following a pre-planned interim analysis, Part B of the study was closed to enrolment after 17 subjects had completed the study.
Groups:
- Part A (0.8 mg/kg; 1.2 mg/kg; 1.8 mg/kg); Part A (0.8 mg/kg; 1.2 mg/kg; Placebo); Part A (0.8 mg/kg; Placebo; 1.8 mg/kg); Part A (Placebo; 1.2 mg/kg; 1.8 mg/kg): Doses were administered as a single intravenous infusion on Days 1, 4 and 7
- Part B, LAT8881/Placebo: LAT8881 was given as a single intravenous infusion on Day 1 at a dose of 1.8 mg/kg. Placebo was administered as a single intravenous infusion on the following day
- Part B Placebo/LAT8881: Placebo was administered as a single intravenous infusion on Day 1. LAT8881 was given as a single intravenous infusion on the following day at a dose of 1.8 mg/kg
Period: Overall Study
Arm/Group | Part A (0.8 mg/kg; 1.2 mg/kg; 1.8 mg/kg) | Part A (0.8 mg/kg; 1.2 mg/kg; Placebo) | Part A (0.8 mg/kg; Placebo; 1.8 mg/kg) | Part A (Placebo; 1.2 mg/kg; 1.8 mg/kg) | Part B, LAT8881/Placebo | Part B Placebo/LAT8881
Started | 2 | 2 | 2 | 3 (One subject withdrew before commencement of treatment) | 8 | 9
Completed | 2 | 2 | 2 | 2 | 8 | 9
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A (0.8 mg/kg; 1.2 mg/kg; 1.8 mg/kg) | Part A (0.8 mg/kg; 1.2 mg/kg; Placebo) | Part A (0.8 mg/kg; Placebo; 1.8 mg/kg) | Part A (Placebo; 1.2 mg/kg; 1.8 mg/kg) | Part B, LAT8881/Placebo | Part B Placebo/LAT8881 | Total
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 8 | 9 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (4.2) | 28.5 (3.5) | 21.0 (1.4) | 26.0 (4.0) | 51.9 (13.5) | 56.0 (11.9) | 44.2 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 1 | 3 | 6 | 15
  Male | 0 | 0 | 1 | 2 | 5 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 2 | 2 | 3 | 7 | 9 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 2 | 2 | 2 | 3 | 8 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Adverse Events by Dose (Part A)
Description: The number of participants in Part A with the following adverse events will be reported by dose (with all placebo subjects combined)
  * All adverse events
  * Serious adverse events
  * Adverse events leading to premature discontinuation of Investigational Medicinal Product (IMP)
  * Adverse events by intensity
  * Adverse events by relationship to IMP
Time Frame: From first dose of LAT8881 to end of study visit (Day 14)
Population: Safety population. This population included all subjects who received at least one dose of IMP and had at least one post dose safety assessment.
Measure: Number; unit: participants
Groups:
- Part A, LAT8881 0.8 mg/kg: LAT8881 was given as a single intravenous infusion at a dose of 0.8 mg/kg
- Part A, LAT8881 1.2 mg/kg: LAT8881 was given as a single intravenous infusion at a dose of 1.2 mg/kg
- Part A, LAT8881 1.8 mg/kg: LAT8881 was given as a single intravenous infusion at a dose of 1.8 mg/kg
- Part A, Placebo: Placebo was given as a single intravenous infusion
Arm/Group | Part A, LAT8881 0.8 mg/kg | Part A, LAT8881 1.2 mg/kg | Part A, LAT8881 1.8 mg/kg | Part A, Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
participants
  Any adverse event | 1 | 1 | 2 | 2
  Serious adverse event | 0 | 0 | 0 | 0
  Adverse events leading to premature discontinuation of Investigational Medicinal Product (IMP) | 0 | 0 | 0 | 0
  Adverse event of Grade 3 or 4 severity | 0 | 0 | 0 | 0
  Adverse events related to IMP (possibly, probably or definitely) | 0 | 0 | 2 | 1

2. Primary Outcome: Change in Baseline Pain With Intravenous LAT8881 in Patients With Lumbar Radicular Pain (Part B)
Description: Change in pain from baseline is measured on on a 0-10 Visual Analogue Scale (VAS). The VAS consists of a 10 cm line with two endpoints representing 0 (no pain) and 10 (pain as bad as it could possibly be). The subject is asked to rate their current level of pain by placing a mark on the line and the distance from 0 is measured to provide a pain intensity score out of 10.
  VAS measurements are taken as the infusion starts and at 15 minute intervals for the first hour, then every thirty minutes for an additional two hours, then hourly until 6 hours from infusion commencement
Time Frame: From start of infusion to 6 hours after start of infusion
Population: Full Analysis Set. This population included all enrolled and randomised participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- LAT8881: LAT8881 was given as a single intravenous infusion at a dose of 1.8 mg/kg.
- Placebo: Matching placebo'was given as a single intravenous infusion.
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 17 | 17
score on a scale
  Pre-dose VAS score | 3.7 (2.7) | 3.1 (2.3)
  Change from pre-dose score at 0.25 hours: number analyzed (Participants) | 16 | 17
  Change from pre-dose score at 0.25 hours | -0.8 (1.8) | -0.3 (1.1)
  Change from pre-dose score at 0.5 hours | -0.8 (2.0) | -0.3 (1.5)
  Change from pre-dose score at 0.75 hours | -1.0 (1.8) | -0.5 (1.5)
  Change from pre-dose score at 1.0 hours | -1.1 (2.2) | -0.6 (1.4)
  Change from pre-dose score at 1.5 hours | -0.8 (1.8) | -0.5 (1.1)
  Change from pre-dose score at 2 hours | -0.8 (2.0) | -0.4 (1.4)
  Change from pre-dose score at 2.5 hours | -0.8 (2.1) | -0.6 (1.4)
  Change from pre-dose score at 3 hours | -0.6 (1.9) | -0.7 (1.5)
  Change from pre-dose score at 3.5 hours | -0.8 (2.1) | -0.8 (1.4)
  Change from pre-dose score at 4 hours | -0.9 (2.0) | -0.5 (1.5)
  Change from pre-dose score at 5 hours | -1.0 (2.2) | -0.7 (1.6)
  Change from pre-dose score at 6 hours | -1.2 (2.0) | -0.8 (1.4)
Statistical Analysis 1: Comparison: LAT8881 vs Placebo; Change from baseline VAS score at 0.25 hours; Test type: Superiority — No formal sample size estimation was undertaken due to the exploratory nature of the study. Analysis was based a mixed model repeated measures model, with fixed-effects including treatment, time point and period factors. Baseline was included as a covariate. Random effects for participants and participant by period were also included; p = 0.5196, Mixed Models Analysis — No adjustment for multiple comparisons was made due to the exploratory nature of the study; Mean Difference (Net) = -0.25, 95% CI 2-sided [-1.02 to 0.52] — Difference is LAT8881 minus placebo
Statistical Analysis 2: Comparison: LAT8881 vs Placebo; Change in VAS score from baseline at 0.5 hours; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.3983, Mixed Models Analysis — No adjustment for multiple comparisons has been made due to the exploratory nature of the study; Mean Difference (Net) = -0.32, 95% CI 2-sided [-1.09 to 0.44] — Difference is LAT8881 minus placebo
Statistical Analysis 3: Comparison: LAT8881 vs Placebo; Change from baseline VAS score at 0.75 hours; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.4890, Mixed Models Analysis — No adjustment for multiple comparisons was made due to the exploratory nature of the study; Mean Difference (Net) = -0.26, 95% CI 2-sided [-1.03 to 0.5] — Difference is LAT8881 minus placebo
Statistical Analysis 4: Comparison: LAT8881 vs Placebo; Change from baseline VAS score at 1 hour; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.5903, Mixed Models Analysis — No adjustment for multiple comparisons was made due to the exploratory nature of the study; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.97 to 0.56] — Difference is LAT8881 minus placebo
Statistical Analysis 5: Comparison: LAT8881 vs Placebo; Change from baseline VAS score at 1.5 hours; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.7352, Mixed Models Analysis — No adjustment for multiple comparisons was made due to the exploratory nature of the study; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.90 to 0.64] — Difference is LAT8881 minus placebo
Statistical Analysis 6: Comparison: LAT8881 vs Placebo; Change from baseline VAS score at 2 hours; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.6892, Mixed Models Analysis — No adjustment for multiple comparisons was made due to the exploratory nature of the study; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.92 to 0.61] — Difference is LAT8881 minus placebo
Statistical Analysis 7: Comparison: LAT8881 vs Placebo; Change from baseline VAS score at 2.5 hours; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.9767, Mixed Models Analysis — No adjustment for multiple comparisons was made due to the exploratory nature of the study; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.78 to 0.76] — Difference is LAT8881 minus placebo
Statistical Analysis 8: Comparison: LAT8881 vs Placebo; Change from baseline VAS score at 3 hours; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.3964, Mixed Models Analysis — No adjustment for multiple comparisons was made due to the exploratory nature of the study; Median Difference (Net) = 0.32, 95% CI 2-sided [-0.44 to 1.09] — Difference is LAT8881 minus placebo
Statistical Analysis 9: Comparison: LAT8881 vs Placebo; Change from baseline VAS score at 3.5 hours; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.5669, Mixed Models Analysis — No adjustment for multiple comparisons was made due to the exploratory nature of the study; Mean Difference (Net) = 0.22, 95% CI 2-sided [-0.55 to 0.98] — Difference is LAT8881 minus placebo
Statistical Analysis 10: Comparison: LAT8881 vs Placebo; Change from baseline VAS score at 4 hours; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.7006, Mixed Models Analysis — No adjustment for multiple comparisons was made due to the exploratory nature of the study; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.91 to 0.62] — Difference is LAT8881 minus placebo
Statistical Analysis 11: Comparison: LAT8881 vs Placebo; Change from baseline VAS score at 5 hours; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.7940, Mixed Models Analysis — No adjustment for multiple comparisons was made due to the exploratory nature of the study; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.87 to 0.67] — Difference is LAT8881 minus placebo
Statistical Analysis 12: Comparison: LAT8881 vs Placebo; Change from baseline VAS score at 6 hours; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.6892, Mixed Models Analysis; No adjustment for multiple comparisons was made due to the exploratory nature of the study; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.92 to 0.61]; Difference is LAT8881 minus placebo

3. Secondary Outcome: Maximum Plasma LAT8881 Concentration (Cmax) After Intravenous LAT8881 (Part A)
Description: LAT8881 is measured in plasma samples taken pre-dose and at 5 minutes, 0.25, 0.5, 1, 2, 4 and 6 hours after IMP administration
Time Frame: Up to 6 hours after the start of each infusion
Population: Subgroup of the pharmacokinetic population. Data for subjects with no measurable levels of LAT8881 were excluded from the summary.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A, LAT8881 0.8 mg/kg | Part A, LAT8881 1.2 mg/kg | Part A, LAT8881 1.8 mg/kg | Part A, Placebo
Number analyzed (Participants) | 3 | 5 | 5 | 0
ng/mL | 12.6 (19.1) | 10.2 (12.9) | 13.8 (14.1) |

4. Secondary Outcome: Time to Maximum Plasma LAT8881 Concentration (Tmax) After Intravenous LAT8881 (Part A)
Description: LAT8881 was measured in plasma samples taken pre-dose and at 5 minutes, 0.25, 0.5, 1, 2, 4 and 6 hours after IMP administration
Time Frame: Up to 6 hours after the start of each infusion
Population: Subgroup of the pharmacokinetic population. Data for a subject with no measurable levels of LAT8881 were excluded from the summary.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A, LAT8881 0.8 mg/kg | Part A, LAT8881 1.2 mg/kg | Part A, LAT8881 1.8 mg/kg | Part A, Placebo
Number analyzed (Participants) | 3 | 5 | 5 | 0
hours | 0.08 (0) | 0.08 (0) | 0.08 (0) |

5. Secondary Outcome: Area Under the Concentration Time Curve From Zero to Infinity (AUC0-inf) After Intravenous LAT8881 (Part A)
Description: LAT8881 was measured in plasma samples taken pre-dose and at 5 minutes, 0.25, 0.5, 1, 2, 4 and 6 hours after IMP administration. (AUC0-inf) was calculated only if there were at least three quantifiable data points.
Time Frame: Up to 6 hours after the start of each infusion
Population: Subgroup of the pharmacokinetic population. Data for subjects with no measurable levels of LAT8881 were excluded from the summary. (AUC0-inf) was not calculated as the criteria of at least three quantifiable data points was not met
Measure: Mean (Standard Deviation); unit: ng/mL*h
Arm/Group | Part A, LAT8881 0.8 mg/kg | Part A, LAT8881 1.2 mg/kg | Part A, LAT8881 1.8 mg/kg | Part A, Placebo
Number analyzed (Participants) | 3 | 5 | 5 | 0
ng/mL*h | NA (NA) — (AUC0-inf) was not calculated as the criteria of at least three quantifiable data points was not met | NA (NA) — (AUC0-inf) was not calculated as the criteria of at least three quantifiable data points was not met | NA (NA) — (AUC0-inf) was not calculated as the criteria of at least three quantifiable data points was not met |

6. Secondary Outcome: Terminal Elimination Half Life (T1/2), (Part A)
Description: LAT8881 was measured in plasma samples taken pre-dose and at 5 minutes, 0.25, 0.5, 1, 2, 4 and 6 hours after IMP administration. The terminal elimination half life was only determined if there were at least three quantifiable elimination phase data points.
Time Frame: Up to 6 hours after the start of each infusion
Population: Subgroup of the pharmacokinetic population. Data for a subject with no measurable levels of LAT8881 were excluded from the summary. Terminal half-life could not be determined as the criteria of at least three quantifiable elimination phase data points was not met
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A, LAT8881 0.8 mg/kg | Part A, LAT8881 1.2 mg/kg | Part A, LAT8881 1.8 mg/kg | Part A, Placebo
Number analyzed (Participants) | 3 | 5 | 5 | 0
hours | NA (NA) — Terminal half-life could not be determined as the criteria of at least three quantifiable elimination phase data points was not met | NA (NA) — Terminal half-life could not be determined as the criteria of at least three quantifiable elimination phase data points was not met | NA (NA) — Terminal half-life could not be determined as the criteria of at least three quantifiable elimination phase data points was not met |

7. Secondary Outcome: Patient General Impression of Change (Part B)
Description: The Patient General Impression of Change (PGIC) is a single-item rating by subjects of their improvement with treatment during a clinical trial. Participants were asked to select one of the following options after each treatment: very much improved, much improved, slightly improved, no change, slightly worse, much worse, very much worse.
Time Frame: 6 hours after the start of each infusion
Population: PGIC was measured in the Full Analysis Set. This population consisted of all subjects who were enrolled and randomised into the study
Measure: Count of Participants; unit: Participants
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 17 | 17
Participants
  Very much improved | 2 | 0
  Much improved | 3 | 2
  Slightly improved | 4 | 11
  No change | 7 | 4
  Slightly worse | 1 | 0
  Much worse | 0 | 0
  Very much worse | 0 | 0

8. Secondary Outcome: The Number of Participants With Adverse Events After Intravenous LAT8881 in Patients With Lumbar Radicular Pain (Part B)
Description: The number of participants in Part B with the following adverse events will be reported after placebo and after intravenous LAT8881
  * All adverse events
  * Serious adverse events
  * Adverse events leading to premature discontinuation of Investigational Medicinal Product (IMP)
  * Adverse events by intensity
  * Adverse events by relationship to IMP
Time Frame: From start of infusion to end of study visit (Day 9)
Population: The safety population consisted of all randomized participants who received at least one dose of IMP and had at least one post dose safety assessment.
Measure: Number; unit: participants
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 17 | 17
participants
  Any adverse event | 5 | 4
  Serious adverse event | 0 | 0
  Adverse event leading to discontinuation | 0 | 0
  Adverse event of Grade 3 or 4 severity | 0 | 0

9. Other Pre Specified Outcome: The Effect of LAT8881, Compared With Placebo, on VAS Pain Scores During a Straight-leg Nerve Stretch.
Description: Change in pain from baseline is measured on a 0-10 Visual Analogue Scale (VAS). The VAS consists of a 10 cm line with two endpoints representing 0 (no pain) and 10 (pain as bad as it could possibly be). The subject is asked to rate their current level of pain on leg raising by placing a mark on the line and the distance from 0 is measured to provide a pain intensity score out of 10. VAS measurements are taken as the infusion starts and at 15 minute intervals for the first hour, then every thirty minutes for an additional two hours, then hourly until 6 hours from infusion commencement.
  Each measurement ranges from 0 to 10. The difference from the pre-dose score is calculated at specified timepoints up to 6 hours post-dose.
Time Frame: From start of infusion to 6 hours after start of infusion
Population: Full analysis set. This population included all subjects who were enrolled and randomised into the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LAT8881 | Placebo
Number analyzed (Participants) | 17 | 17
score on a scale
  Pre-dose VAS score | 5.2 (2.6) | 4.8 (2.4)
  VAS change from baseline at 0.25 hours | -0.3 (1.7) | 0.2 (0.9)
  VAS change from baseline at 0.5 hours | -0.8 (1.2) | -0.3 (1.3)
  VAS change from baseline at 0.75 hours | -1.1 (1.4) | -0.2 (1.5)
  VAS change from baseline at 1 hour | -1.1 (1.7) | -0.2 (1.5)
  VAS change from baseline at 1.5 hours | -1.2 (1.9) | 0.0 (1.5)
  VAS change from baseline at 2 hours | -0.9 (1.9) | -0.3 (1.5)
  VAS change from baseline at 2.5 hours | -1.0 (1.9) | -0.1 (1.6)
  VAS change from baseline at 3 hours | -1.1 (1.9) | -0.4 (1.7)
  VAS change from baseline at 3.5 hours | -1.3 (2.1) | -0.4 (1.7)
  VAS change from baseline at 4 hours | -1.3 (2.6) | -0.6 (2.2)
  VAS change from baseline at 5 hours | -1.6 (2.2) | -0.7 (2.0)
  VAS change from baseline at 6 hours | -1.3 (2.1) | -1.2 (2.2)

ADVERSE EVENTS:
Time Frame: All events occurring during and following the first administration of IMP were reported as adverse events until the completion of the End of Study Evaluation visit (Day 14 for Part A, Day 9 for Part B).
Groups:
- Part B, LAT8881: LAT8881 was given as a single intravenous infusion at a dose of 1.8 mg/kg
- Part B, Placebo: Placebo was given as a single intravenous infusion
Arm/Group | Part A, LAT8881 0.8 mg/kg | Part A, LAT8881 1.2 mg/kg | Part A, LAT8881 1.8 mg/kg | Part A, Placebo | Part B, LAT8881 | Part B, Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 2/6 | 2/6 | 5/17 | 4/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A, LAT8881 0.8 mg/kg (N=6) | Part A, LAT8881 1.2 mg/kg (N=6) | Part A, LAT8881 1.8 mg/kg (N=6) | Part A, Placebo (N=6) | Part B, LAT8881 (N=17) | Part B, Placebo (N=17)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachyardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphoria (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reflex gastritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Every participating investigator agrees to keep all information and results concerning the study and the investigational product confidential for as long as the data remain unpublished.

DOCUMENTS (2):
  • Study Protocol (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT05298306/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT05298306/SAP_001.pdf